CLINICAL TRIAL: NCT03271086
Title: Family Centered Relaxation Breathing Training in the Pediatrics Outpatient Clinic
Brief Title: Relaxation Breathing Training for Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never started.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-36659
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Stress Disorder; Biofeedback
Keywords: Relaxation training; Pediatric clinic; Children 6-11 years; Text messaging
MeSH Terms: conditions — Stress Disorders, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation breathing training (Experimental): Dyads of a parent and their child in this group will receive training on how to use breathing to relax with the StressEraser in the pediatric clinic and will then practice the breathing for about 4 weeks They will also complete a baseline questionnaire and two questionnaires one month after the training.
  Interventions: Behavioral: The StressEraser
- Technology-enhanced relaxation breathing (Experimental): Dyads of a parent and their child in this group will receive technology-enhanced training on how to use breathing to relax with the StressEraser and the app Breathe2Relax in the pediatric clinic and will then practice the breathing for about 4 weeks and weekly receive weekly reminder text messages to practice their relaxation breathing. They will also complete a baseline questionnaire and two questionnaires one month after the training.
  Interventions: Behavioral: The StressEraser; Behavioral: Breathe2Relax; Behavioral: Reminder text messages

INTERVENTIONS:
Behavioral: The StressEraser — The StressEraser is a handheld biofeedback device that measures heart rate variability (HRV). Heart rate increases during inspiration and decreases during expiration. The HRV, depicted on a miniature screen, essentially represents respirations. The investigator's prior study demonstrated that the device is easily mastered and acceptable to children above 6 years of age.
Behavioral: Breathe2Relax — Breathe2Relax is a free mobile app, developed by the Dept. of Defense's National Center for Telehealth and Technology to help veterans with PTSD and others use breathing practice for stress management. This application guides users in relaxation breathing and is available for both android and iOS phones. It is adapted for children 6 years and up. For instance, the cycles can be shortened for children, there is a selection of quiet music and the user can choose backgrounds for personalization.
  Arms: Technology-enhanced relaxation breathing
Behavioral: Reminder text messages — Weekly texts will be sent out to parents in the technology-enhanced relaxation breathing group to as reminders to practice the daily relaxation breathing with their child.
  Arms: Technology-enhanced relaxation breathing

SUMMARY:
Family-centered Relaxation Breathing Training in the Pediatric Outpatient Clinic:

The long term goal is to apply simple, low cost, assistive technologies (heart rate variability [HRV] biofeedback together with mobile health tools) to teach relaxation breathing in the Boston Medical Center pediatric clinic setting following a trauma-informed care model. For this research both a mobile app for relaxation breathing skills and reminder text messages will be provided for the at-risk target population. The investigators will assess the feasibility and acceptability of relaxation breathing intervention in 60 parent-child dyads. These dyads will be randomly assigned to receive either (1) biofeedback relaxation training alone or (2) Technology-enhanced relaxation breathing (biofeedback relaxation training together with mobile health tools). Outcome measures will assess relaxation breathing practice, anxiety, and parental stress at the time of the intervention and at one month follow up.

DETAILED DESCRIPTION:
After consent is signed, a baseline questionnaire will be given to the participant, including demographics and baseline data followed by randomization into one of the following groups:Relaxation breathing training alone or Technology-enhanced relaxation breathing.The intervention will occur through the use of the StressEraser, Breathe2Relax and text messaging.

1. The StressEraser is a handheld biofeedback device that measures heart rate variability (HRV). Heart rate increases during inspiration and decreases during expiration. This HRV, depicted on a miniature screen, essentially represents respirations. We have been using this device in the pediatric outpatient department over the past two years (in a non research entity) and it has been well accepted by children 6 years of age and above. In our prior study, which took place in school, the device was also easily mastered and acceptable to children above 6 years of age.
2. Breathe2Relax is a free mobile app, developed by the Dept. of Defense's National Center for Telehealth and Technology to help veterans with PTSD and others use breathing practice for stress management. This application guides users in relaxation breathing and is available for both android and iOS phones. It is adapted for children 6 years and up. The user downloads the app. and is walked through steps that easily explain the purpose of the app (to guide relaxation breathing). The active part of the app shows a tube that fills in during inspiration and empties during expiration. For children the cycle lengths can be shortened which is explained to participating parents by the research team. There is a selection of quiet music and the user can choose backgrounds for personalization. The Breath2Relax app will be downloaded for the RT-enhanced group at the time of the intervention for the RT-enhanced group, and the parent will be shown how to modify the length of the breath cycle depending on their child's age.
3. Text messages: Weekly texts will be sent out to parents in the RT-enhanced group regarding relaxation breathing and to remind parents to practice the daily relaxation breathing with their child.

For the breathing training, the study research assistant (RA) will follow the standardized protocol used in BMC pediatric clinic over the past two years. The child is taught firstand learns how to use relaxation breathing and then the child teaches their parent how it works with the support of the RA. This step assures that the child has learned the relaxation breathing skills and also creates a moment when relaxation breathing is practiced together by the dyad. The parent-child dyad are encouraged to practice relaxation breathing once daily.Caregivers usually choose bedtime to practice breathing because the practice can be done while the child is in bed.

The training is followed for the Technology-enhanced relaxation breathing group by downloading the Breath2Relax app on the parent's smartphone. Parents will be prompted by the RA to choose a specific time each day to practice the relaxation breathing with their child, and for the Technology-enhanced relaxation breathing group using the Breath2Relax app.

ELIGIBILITY:
Inclusion Criteria:

* child between 6 and 11 years of age and their parent
* primary language either English or Spanish
* parent has a working smartphone

Exclusion Criteria:

* a child who is in Department of Children and Families (DCF) custody whose caregiver is a foster parent
* parent who does not speak or read English or Spanish

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Fidelity to daily relaxation breathing | daily for 4 weeks
  Fidelity to the daily relaxation breathing will be captured from information recorded by the parent in a dairy this will be provided at the end of the relaxation training. They will be instructed to record the number of times daily that they and their child do the relaxation breathing exercises. Data will be entered by the research team 4 weeks post training and the number of times/total number of days post training for each parent and child will be calculated.

SECONDARY OUTCOMES:
Parenting Stress Index Short Form (PSI-SF) | one month follow up
  The PSI-SF is a questionnaire that contains 36 statements written at a 5th-grade reading level, for parents of children 12 years and younger. The PSI/SF yields a Total Stress score from three scales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. The total score is read from percentiles and the 16th - 84th Percentile = Normal range, 85th - 89th Percentile = High range, 90th Percentile or higher = Clinically significant range for parental stress.
Spence Children's Anxiety Scale (SCAS) | one month follow up
  SCAS is a 39 item instrument completed by the parent but only the first 38 items are scored.The parent selects one of the following four responses to the first 38 items: never=0, sometimes=1, often=2, or always=3. Scores can range from 0 to 114 and the higher the score the more anxiety the child has. The 39th item asks the parent if their child is afraid of anything else with a yes or no response; it is not scored..

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Steiner, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No